CLINICAL TRIAL: NCT01143675
Title: The Influence of Local Bone Status on Complications After Surgical Treatment of Proximal Humerus Fractures
Brief Title: Influence of Local Bone Status on Complications After Surgical Treatment of Proximal Humerus Fractures
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FFOB-Hum
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Proximal Humeral Fractures; Poor Bone Quality; Treatment Complications
Keywords: Humerus fractures; Tomography, x-ray computed; Bone and bones; Orthopedic fixation devices; Surgery; Postoperative complications; Osteoporosis; Intraoperative complications; Bone density; Radiography, dual-energy scanned projection
MeSH Terms: conditions — Shoulder Fractures; Humeral Fractures; Postoperative Complications; Osteoporosis; Intraoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate if poor bone quality increases the risk of specific types of treatment complications in patients with proximal humerus fractures treated with open reduction and angle-stable plates (Proximal Humeral Internal Locking System - PHILOS).

DETAILED DESCRIPTION:
More than 70% of patients with a proximal humerus fracture are older than 60 years, up to three quarters are women and the incidence of low-energy fractures increases exponentially with age. The standard diagnostic method for classifying osteoporosis is the measurement of Bone Mineral Density at specific body sites - hip, vertebra or distal radius. Despite the fact that osteoporotic fractures are very frequent at the shoulder, no study investigated the correlation between local bone quality and fracture treatment at the proximal humerus.

There is a concern among the clinicians that osteoporotic bone in proximal humerus fractures increases the risk of treatment complications. However, to our knowledge this has not yet been evaluated in clinical studies. One major reason for this lack of studies is the fact that no standardized method exists for the determination of bone density at the proximal humerus.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed closed fracture (within 10 days) of the proximal humerus
* All dislocated (mod. Neer) proximal humerus fractures except dislocated fractures of the greater and lesser tuberosity
* Primary fracture treatment with a PHILOS-plate
* Age equal greater than 50 and equal younger than 90 years
* Normal function of both shoulders (pre-trauma) according to age
* Monotrauma
* Willing and able to give written informed consent to participate in the study
* Willing and able to participate in the study follow-ups according to the CIP
* Willing and able to comply with the postoperative management program
* Able to understand and read country national language

Exclusion Criteria:

* Open proximal humerus fractures
* Concomitant contralateral proximal humerus fracture
* Previous proximal humerus fracture on either side after the age of 25
* Time to operation > 10 days
* Polytrauma
* Cuff-arthropathy of the contralateral proximal humerus
* Associated nerve or vessel injury
* Regular systemic therapy with corticosteroids due to chronic disease
* Legal incompetence
* Patient received radio- or chemotherapy prior to, during or within the last year
* Currently active cancer
* Recent history of substance abuse (i.e. recreational drugs, alcohol)
* Prisoner
* Currently involved in a pharmaceutical clinical study§
* Has a disease process that would preclude accurate evaluation (e.g. neuromuscular or rheumatic disease, significant psychiatric or metabolic disorders)
* Simultaneous participation in another orthopedic/surgical study with the same or another fracture has to be approved by the AOCID.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic and trauma clinics
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Local bone quality-related complication | From enrollment to 12 months postoperative
  The qualifying events are those involving either directly the local bone and fracture or the implant and its surgical application whether they are anticipated or not.

SECONDARY OUTCOMES:
Bone mineral density at the distal radius by DXA | until 6 week postoperative
  The BMD at the distal radius will be measured by DXA. It will comprise BMD and BMC of the contralateral side. The absolute values for BMD and BMC will be provided as well as the deviations to the T-score according to the manufacturer's reference collective.
Occurence of any complication | 6 weeks
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation.
Occurence of any complication | 3 months
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation.
Occurence of any complication | 12 months
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation.
Range of motion | 6 weeks
  The bilateral range of motion will be measured by clinical examination as follows:
  * Flexion / extension
  * Abduction
  * External / internal rotation
Range of motion | 3 months
  The bilateral range of motion will be measured by clinical examination as follows (110):
  * Flexion / extension
  * Abduction
  * External / internal rotation
Range of motion | at 12 month follow-up
  The bilateral range of motion will be measured by clinical examination as follows (110):
  * Flexion / extension
  * Abduction
  * External / internal rotation
Constant-Murley Score | 3 months
  Functional assessment of shoulder . The range of total scores is 1 to 100 and is composed of a subjective (mainly pain) and an objective parameters.
Constant-Murley Score | 6 weeks
  Functional assessment of shoulder . The range of total scores is 1 to 100 and is composed of a subjective (mainly pain) and an objective parameters.
Constant-Murley Score | 12 months
  Functional assessment of shoulder . The range of total scores is 1 to 100 and is composed of a subjective (mainly pain) and an objective parameters.
Patient self-assessment of shoulder function - SPADI | Baseline
  SPADI assesses the pain and disability associated with shoulder pathology. It is a self-reported index consisting of 13 items divided into two subscales: pain and disability. The range of total scores is 1 to 100.
Patient self-assessment of shoulder function - SPADI | 6 weeks
  SPADI assesses the pain and disability associated with shoulder pathology. It is a self-reported index consisting of 13 items divided into two subscales: pain and disability. The range of total scores is 1 to 100.
Patient self-assessment of shoulder function - SPADI | 3 months
  SPADI assesses the pain and disability associated with shoulder pathology. It is a self-reported index consisting of 13 items divided into two subscales: pain and disability. The range of total scores is 1 to 100.
Patient self-assessment of shoulder function with the SPADI | 6 months
  SPADI assesses the pain and disability associated with shoulder pathology. It is a self-reported index consisting of 13 items divided into two subscales: pain and disability. The range of total scores is 1 to 100.
Patient self-assessment of shoulder function with the SPADI | 12 months
  SPADI assesses the pain and disability associated with shoulder pathology. It is a self-reported index consisting of 13 items divided into two subscales: pain and disability. The range of total scores is 1 to 100.
Disability of the shoulder and hand - DASH | Baseline
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Patient self-assessment of upper extremity function with the DASH | 6 weeks
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Patient self-assessment of upper extremity function with the DASH | 3 months
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Patient self-assessment of upper extremity function with the DASH | 12 months
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Health-related quality of life - EuroQoL5 | Baseline
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
EuroQoL5 | 6 weeks
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
EuroQoL5 | 3 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
EuroQoL5 | 6 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
EuroQoL5 | 12 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
Validation of a Computed Tomography (CT)-based method for BMD-measurement at the proximal humerus | preoperative
  The BMD (mg/cm3) at the proximal humerus will be determined preoperatively for the contralateral side of the fracture with a general purpose CT scanner, according to the protocol. Briefly, a CT of the contralateral humerus is performed measuring simultaneously the European Forearm Phantom (EFP) applied on the patient's midthorax. The measured CT Hounsfield Units (HU) of user-defined ROIs can then be quantified with the EFPbased calibration curve, resulting in BMD-values.
Association between the BMD at the proximal humerus (measured by CT) and the BMD at the distal radius (measured by DXA) | until 6 weeks postoperative
  Bone density measurements at the left and right proximal and distal humerus have been correlated by Diederichs and colleagues. BMD comparison between left and right humeri revealed higher correlations for the distal (R2 = 0.9) and the proximal humerus (R2 = 0.74) than comparison between proximal and distal humerus (R2 = 0.4) (97). These date suggest that the contralateral should be favored to the ipsilateral location when estimating the bone density of a fractured site.
Occurence of any complication | Baseline
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation. The reported complication will be classified by AOCID as either serious or non-serious AE or as an anticipated complication.

CONTACTS AND LOCATIONS:
Overall Officials: Franz Kralinger, MD, Principal Investigator — Medizinische Uni Innsbruck
Locations (10):
- Medizinische Uni Innsbruck, Innsbruck, Tyrol, Austria
- Queen Mary Hospital, Hong Kong, China
- Germany (3):
  - Klinikum rechts der Isar der TU München, Munich, Bavaria
  - Ev. Diakoniewerk Friederikenstift, Hanover, Lower Saxony
  - Campus Virchow-Klinikum, Charité, Berlin
- Switzerland (5):
  - Centre Hosp Univ Vaudois, Lausanne, Canton of Vaud
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Universitätsspital Basel, Basel
  - Kantonsspital, Lucerne
  - Stadtspital Triemli, Zurich

REFERENCES:
- [Derived] Goldhahn S, Kralinger F, Rikli D, Marent M, Goldhahn J. Does osteoporosis increase complication risk in surgical fracture treatment? A protocol combining new endpoints for two prospective multicentre open cohort studies. BMC Musculoskelet Disord. 2010 Nov 9;11:256. doi: 10.1186/1471-2474-11-256. PMID 21062463
- See also: Non profit organization dedicated to improving the care of patients with musculoskeletal injuries and their sequelae through research, development, education and quality assurance in the principles, practice, and result of fracture treatment. — http://www.aofoundation.org